CLINICAL TRIAL: NCT05557656
Title: A Real World Study of Regogfinib in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Real World Study of Regogfinib in HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Collaborators: The Central Hospital of Lishui City (Other); Anhui Provincial Hospital (Other Government); Zhejiang University (Other); Sun Yat-sen University (Other); Wuxi People's Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); ZhuHai Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor, Zhongda Hospital
Other Study IDs: V1.0 20220518
Record Dates: First submitted 2022-09-17; First posted 2022-09-28 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Regorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC participants who received the treatment of Regorafenib: HCC participants who received the treatment of Regorafenib
  Interventions: Drug: Regorafenib 40 MG

INTERVENTIONS:
Drug: Regorafenib 40 MG — participants who received the treatment of Regorafenib
  Other Names: Regorafenib

SUMMARY:
This is a non-interventional observational study with the primary objective of assessing the efficacy of regorafenib in patients with immediate or advanced stage HCC.

DETAILED DESCRIPTION:
1. Study Objectives Primary Objective: To assess the efficacy of regorafenib in patients with immediate or advanced stage HCC Secondary objective: To assess the safety of regorafenib in patients with immediate or advanced stage HCC
2. Study Design This is a multicenter, retrospective, real-world study that will collect data from patients treated with regorafenib at medical centers in China.
3. Data Collection 3.1 Screening Period

The study procedures to be performed at screening include:

1. . Determine eligible subjects according to the inclusion/exclusion criteria and document the results.
2. . Collect demographic characteristics (eg, age, sex, weight, BMI, and ECOG score);
3. . Collect past medical history;
4. . Collect primary tumor site;
5. . Collect information on prior treatments: all treatments received since diagnosis of advanced HCC, including each treatment regimen (including first-line therapy), start and end date, duration, best response;
6. . Collect information on liver function and ECOG score prior to the first dose of regorafenib;
7. . Collect results of laboratory tests performed prior to and after the first dose of regorafenib, including haematology, biochemistry and genetic testing (if any);
8. . Collect imaging data: the last imaging procedure performed prior to the first dose of regorafenib, such as CT, PET-CT, MRI, and whole-body bone scan (with at least 1 measurable lesion); and information related to metastases (such as metastases to lymph node, bone and/or lung).

3.2 Data Review Period of Regorafenib Treatment

The following information obtained during each cycle of regorafenib will be collected retrospectively:

1. . Liver function and ECOG score obtained prior to each dose (ie., the first day of each cycle) of regorafenib;
2. . Initial dose of regorafenib;
3. . Timing and method of dose adjustment, and adjusted doses;
4. . Final daily dose of regorafenib;
5. . Best response, time to best response, and number of treatment cycles;
6. . Imaging findings (including metastatic sites) related to response evaluation;
7. . Hematology laboratory tests (related to the underlying disease, tumor progression, and ADR);
8. . Any adverse reaction and corresponding CTCAE grade;
9. . Interrupted or discontinued treatment;
10. . The most recent laboratory tests (or alternative doctor's advice and tests) performed prior to the first day of each treatment cycle, including but not limit to hematology and biochemistry.

3.3 Progression and Survival Data Collection Period

The following information obtained during each cycle of regorafenib will be collected retrospectively:

1. . Time to progression
2. . Pattern of progression
3. . Subsequent treatment regimen, dose, number of cycles, efficacy;
4. . Survival status, time of death or last follow-up.

4. Study Drug Generic name: Regorafenib Tablets Trade name: Stivarga® English name: Regorafenib Tablets

Dosage strength: 40 mg tablet Dosage form: Tablets Description: Oval tablets with pale-pink film coat Label dose and mode of administration: Recommended dosage is 160 mg, once daily for the first 21 days of each 28-day cycle. A minimum dose of 80 mg/day and a maximum dose of 160 mg/day are recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically or clinically confirmed HCC;
2. Patients with Barcelona Clinic Liver Cancer (BCLC) stage B/C;
3. Patients previously treated with regorafenib for at least one 28-day cycle after only one prior systemic therapy.

Exclusion Criteria:

1. Patients with incomplete information that would impact the assessment of primary endpoint;
2. Patients with medical history of other malignant neoplasms.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with immediate or advanced stage HCC who have been treated with regorafenib from January 2018 to December 2021 following only one prior systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-01-05 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time from the start of regorafenib treatment to the date of death from any cause or last follow-up，whichever came first, assessed up to 60 months
  Overall survival was defined as the time from the start of regorafenib treatment to the date of death from any cause or last follow-up

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from the start of regorafenib treatment to the date of the first documentation of disease progression or death from any cause，whichever came first, assessed up to 60 months.
  Progression-free survival was defined as the time from the start of regorafenib treatment to the date of the first documentation of disease progression or death from any cause.
Time to progression (TTP) | Time from the start of regorafenib treatment to the date of the first documentation of disease progression，whichever came first, assessed up to 60 months
  Time to progression was defined as the time from the start of regorafenib treatment to the date of the first documentation of disease progression.
Objective response rate (ORR) | Time from the start of regorafenib treatment to the date of the first documentation of objective response，assessed up to 60 months.
  Objective response rate was defined as the proportion of patients with CR or PR in the overall population
Disease control rate (DCR) | Time from the start of regorafenib treatment to the date of the first documentation of CR or PR or stable，assessed up to 60 months.
  Disease control rate was defined as the proportion of patients with CR or PR or stable disease (SD) in the overall population
Adverse events (AEs) | Time from the start of regorafenib treatment to the date of death or last follow up，whichever came first,assessed up to 60 months.
  adverse events (AEs) (including type and grade according to CTCAE 5.0)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Result] Zheng R, Qu C, Zhang S, Zeng H, Sun K, Gu X, Xia C, Yang Z, Li H, Wei W, Chen W, He J. Liver cancer incidence and mortality in China: Temporal trends and projections to 2030. Chin J Cancer Res. 2018 Dec;30(6):571-579. doi: 10.21147/j.issn.1000-9604.2018.06.01. PMID 30700925
- [Result] Zeng H, Chen W, Zheng R, Zhang S, Ji JS, Zou X, Xia C, Sun K, Yang Z, Li H, Wang N, Han R, Liu S, Li H, Mu H, He Y, Xu Y, Fu Z, Zhou Y, Jiang J, Yang Y, Chen J, Wei K, Fan D, Wang J, Fu F, Zhao D, Song G, Chen J, Jiang C, Zhou X, Gu X, Jin F, Li Q, Li Y, Wu T, Yan C, Dong J, Hua Z, Baade P, Bray F, Jemal A, Yu XQ, He J. Changing cancer survival in China during 2003-15: a pooled analysis of 17 population-based cancer registries. Lancet Glob Health. 2018 May;6(5):e555-e567. doi: 10.1016/S2214-109X(18)30127-X. PMID 29653628
- [Result] Craig AJ, von Felden J, Garcia-Lezana T, Sarcognato S, Villanueva A. Tumour evolution in hepatocellular carcinoma. Nat Rev Gastroenterol Hepatol. 2020 Mar;17(3):139-152. doi: 10.1038/s41575-019-0229-4. Epub 2019 Dec 2. PMID 31792430
- [Result] Kudo M, Trevisani F, Abou-Alfa GK, Rimassa L. Hepatocellular Carcinoma: Therapeutic Guidelines and Medical Treatment. Liver Cancer. 2016 Nov;6(1):16-26. doi: 10.1159/000449343. Epub 2016 Nov 29. PMID 27995084
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Result] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Result] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Result] European Association for Study of Liver; European Organisation for Research and Treatment of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. Eur J Cancer. 2012 Mar;48(5):599-641. doi: 10.1016/j.ejca.2011.12.021. No abstract available. PMID 22424278
- [Result] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Result] Arai H, Battaglin F, Wang J, Lo JH, Soni S, Zhang W, Lenz HJ. Molecular insight of regorafenib treatment for colorectal cancer. Cancer Treat Rev. 2019 Dec;81:101912. doi: 10.1016/j.ctrv.2019.101912. Epub 2019 Oct 28. PMID 31715423
- [Result] Lee MJ, Chang SW, Kim JH, Lee YS, Cho SB, Seo YS, Yim HJ, Hwang SY, Lee HW, Chang Y, Jang JY. Real-world systemic sequential therapy with sorafenib and regorafenib for advanced hepatocellular carcinoma: a multicenter retrospective study in Korea. Invest New Drugs. 2021 Feb;39(1):260-268. doi: 10.1007/s10637-020-00977-4. Epub 2020 Aug 4. PMID 32749658
- [Result] Sung PS, Jang JW, Lee J, Lee SK, Lee HL, Yang H, Nam HC, Lee SW, Bae SH, Choi JY, Han NI, Yoon SK. Real-World Outcomes of Nivolumab in Patients With Unresectable Hepatocellular Carcinoma in an Endemic Area of Hepatitis B Virus Infection. Front Oncol. 2020 Jun 30;10:1043. doi: 10.3389/fonc.2020.01043. eCollection 2020. PMID 32695681
- [Result] Nair A, Reece K, Donoghue MB, Yuan WV, Rodriguez L, Keegan P, Pazdur R. FDA Supplemental Approval Summary: Lenvatinib for the Treatment of Unresectable Hepatocellular Carcinoma. Oncologist. 2021 Mar;26(3):e484-e491. doi: 10.1002/onco.13566. Epub 2020 Nov 10. PMID 33044793
- See also: Related Info — http://gco.iarc.fr/today/data/factsheets/cancers/11-Liver-fact-sheet.pdf